CLINICAL TRIAL: NCT05268614
Title: Risk Adapted De-Intensification of Radio-Chemotherapy for Favorable Prognosis Oropharyngeal Squamous Cell Carcinoma Based on HPV Subtype and Plasma Circulating Free HPV DNA Level and Clearance Rate
Brief Title: Risk Adapted De-Intensification of Radio-Chemotherapy for Oropharyngeal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Naveris, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-HN-004; OCR41015 (Other: University of Florida)
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: Oropharyngeal Squamous Cell Carcinoma; chemo-radiotherapy; cfHPV DNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemo-radiotherapy (Experimental): Participants will receive chemo-radiotherapy.
  Interventions: Radiation: Radiation therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation therapy — Participants will receive either 70 gray (Gy), 60 Gy, or 50 Gy of radiation based on the following criteria:
  70 Gy: Pretreatment level of plasma circulating free HPV DNA (cfHPV DNA) ≤ 12 copies/mL
  60 Gy: Tumor tissue positive for HPV subtype other than 16 OR Pretreatment level of cfHPV DNA 13-99 copies/mL OR Pretreatment level of cfHPV DNA ≥ 100 copies/mL AND <95% decrease in the level cfHPV DNA by the end of week 4 of radiation therapy
  50 Gy: Tumor tissue positive for HPV subtype 16, pretreatment level of cfHPV DNA ≥ 100 copies/mL, AND ≥ 95% decrease in the level cfHPV DNA by the end of week 4 of radiation therapy
Drug: Cisplatin — All participants will receive 40 mg/m2 of cisplatin intravenously over 60 minutes weekly during radiation therapy.
  If cisplatin is not recommended by the treating medical oncologist or is not tolerated, it is permissible to switch to an alternative chemotherapy regimen per institutional practice, but chemotherapy should not be discontinued unless mandated by the patient's condition.

SUMMARY:
This study builds on the results of several prior studies that we have been involved with to test the hypothesis that Risk-Adapted De-Intensification of Radiation Therapy and chemotherapy based on HPV subtype, plasma circulating free HPV DNA (cfHPV DNA) level, and cfHPV DNA clearance rate produces Local-Regional Control rates that are similar to what has been achieved with more aggressive therapy in patients with Favorable Prognosis Oropharyngeal Squamous Cell Carcinoma (OPSCC).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age (no upper age limit)
2. T0-3 ≤4cm, N0 to N2, M0 squamous cell carcinoma of the oropharynx by AJCC 8th Edition staging. If T0 the adenopathy must be predominantly in Level 2.
3. Tissue diagnosis of HPV and/or p16 positivity from the primary site or an associated lymph node.
4. Radiologic confirmation of the absence of lung metastasis within 12 weeks prior to treatment; at a minimum, CT of the chest is required. PET-CT is acceptable.
5. ECOG Performance Status 0-2
6. ≤10 pack-years of smoking or no smoking for ≥ 10 years
7. Eligible for chemotherapy
8. CBC/differential obtained within 12 weeks prior to treatment, with adequate bone marrow function defined as follows:

   * Platelets ≥ 100,000 cells/mm3
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
9. Adequate renal and hepatic function within 12 weeks prior to treatment, defined as follows:

   * Serum creatinine < 2.0 mg/dl
   * Total bilirubin < 2 x the institutional ULN (upper limit of normal)
   * AST or ALT < 3 x the institutional ULN
   * Note that physician attestation of patient having no known history of liver disease can take the place of bilirubin and AST/ALT labs.
10. Negative pregnancy test within 3 weeks prior to treatment for women of childbearing potential.
11. People of childbearing potential (POCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 14 months after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, people of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.

    POCBP includes any person who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:
    * Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
    * For people with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
12. Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 14 months following the last dose of study drug.
13. Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Prior radiotherapy or chemotherapy for this cancer.
2. Prior surgery with curative intent for this OPSCC.
3. Patients who have undergone tonsillectomy for diagnosis or excisional biopsy of a neck node for diagnosis are eligible provided there is "gross" cancer present at the primary site or in the neck at the start of radiation therapy on this protocol with "gross" defined as visible on an imaging study.
4. Prior history of radiation therapy to the head and neck, with the exception of skin cancer treated with a small (≤ 9cm3) field with 6 - 9 MeV electron beam or 50 - 250 kVp photon beam.
5. Prior history of chemotherapy or immunotherapy for cancer within the last 10 years
6. Prior history within 5 years of invasive cancer with the exception of:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin, stage 1-2
   * Prostate cancer without distant metastases (stage M0)
   * Thyroid cancer without distant metastases (stage M0)
7. Prior history of invasive squamous cell carcinoma of a mucosal site in the head or neck treated with surgery alone within the last 5 years.
8. Prior history of invasive malignant melanoma or Merkel cell carcinoma of the head or neck treated with surgery alone in the past 5 years.
9. Inhalation smoking of tobacco within the last 10 years with > 10 pack-year equivalent history.
10. Currently taking Disease Modifying Rheumatoid Drugs (DMRDs) or immunosuppressive medication, for example as for organ transplant or multiple sclerosis.
11. Severe, active co-morbidity, defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    * Transmural myocardial infarction within the last 6 months
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; Note, however, coagulation parameters are not required for entry into this protocol.
    * Evidence of ACTIVE systemic lupus or scleroderma
    * Psoriatic arthritis
12. Known HIV positivity. HIV positive patients are known to have worse clinical outcomes especially for local, regional, and distant cancer control. This poorer prognosis is thought to be secondary to a compromised immune system. Thus, de-intensification of radiation and chemotherapy is not justifiable in this population. HIV testing at the time of enrollment is not required.
13. Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 14 months after the last dose of study drug.
14. People who are pregnant or breastfeeding.
15. Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Local-Regional Control Rate | 2 years
  Determine the Local-Regional Control Rate, defined as the absence of recurrence of OPSCC at the primary site or in a neck node that was included in a radiation therapy target volume

SECONDARY OUTCOMES:
Local Control Rate | 2 years
  Determine the local control rate, defined as as the absence of recurrence of OPSCC at the primary site
Regional Control Rate | 2 years
  Determine the regional control rate, defined as the absence of recurrence in a neck node
Disease-Free Survival | 2 years
  Determine the disease-free survival, defined as the time from the first day of radiation to the date of first recurrence (local, regional, or distant)
Distant Metastasis-Free Survival | 2 years
  Determine the distant metastasis-free survival, defined as the time from the first day of radiation to the date distant metastases are confirmed
Overall Survival | 2 years
  Determine the overall survival, defined as the time from the first day of radiation to the date of death
Participant Quality of Life | 2 years
  Assess participant quality of life using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) instrument. The EORTC QLQ-C30 measures ability to perform everyday activities and whether the subject has experienced select physical symptoms on a scale of 1-4 (with 1 meaning "Not at all" and 4 meaning "Very much"), as well as overall quality of life and overall health over the past week on a scale from 1-7 (with 1 meaning "Very Poor" and 7 meaning "Excellent"). For questions measuring ability to perform everyday activities, overall quality of life, and overall health, a higher score means better functioning, quality of life or overall health. For questions related to symptoms, a higher score means that the subject has experienced that symptom more.
Swallowing Ability | 2 years
  Assess participant swallowing ability using the Eating Assessment Tool (EAT-10) instrument. The EAT-10 instrument asks subjects to rate the extent to which ten scenarios related to swallowing are problematic for them on a scale of 0-4, where a score of 0 means "No Problem" and a score of 4 means "Severe Problem".
Swallowing Ability | 2 years
  Assess participant swallowing ability using the M.D. Anderson Dysphagia Inventory (MDADI) instrument. The MDADI asks participants if they strongly agree, agree, have no opinion, disagree, or strongly disagree with twenty statements related to swallowing. Each response is given a score of 1 to 5 points and all the scores are summed to produce a composite score ranging from 20 to 100, where a higher score means better functioning related to swallowing.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Hitchcock, MD, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - UF Health Proton Therapy Institute, Jacksonville, Florida
  - Medical University of South Carolina, Charleston, South Carolina